CLINICAL TRIAL: NCT02623478
Title: Pharmacokinetics, Glucodynamics, Safety, and Tolerability of a Novel Insulin Lispro Formulation in Patients With Type 1 Diabetes Mellitus on Continuous Subcutaneous Insulin Infusion Therapy
Brief Title: A Study of a Novel Insulin Lispro Formulation in Participants With Type 1 Diabetes Mellitus Using Insulin Pumps
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in clinical strategy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15639; F3Z-FW-ITCD (Other: Eli Lilly and Company); 2015-003353-18 (EudraCT Number)
Record Dates: First submitted 2015-12-03; First posted 2015-12-07 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin Lispro - Test Formulation (Experimental): Novel formulation of insulin lispro delivered via an insulin pump as a continuous infusion under the skin, with intermittent bolus doses during meals for two 3-day periods
  Interventions: Drug: Insulin Lispro
- Insulin Lispro - Reference Formulation (Active Comparator): Marketed formulation of insulin lispro delivered via an insulin pump as a continuous infusion under the skin, with intermittent bolus doses during meals for two 3-day periods
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: Insulin Lispro — Administered subcutaneously (SC)
  Other Names: Humalog

SUMMARY:
This study evaluates a new test formulation of a glucose lowering drug, insulin lispro, delivered by an insulin pump continuously under the skin. The study will be conducted in participants with type 1 diabetes mellitus to investigate how the human body processes the new test formulation and its effect on blood sugar levels when it is delivered via an insulin pump. Side effects and tolerability will be documented. The study will last about 4 to 11 weeks, including screening, lead-in and follow up. Screening is required within 28 days prior to entering the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with Type 1 Diabetes Mellitus (T1DM) who are receiving insulin therapy via an approved insulin pump
* Have a body mass index (BMI) of 18.5 to 33 kilogram per square meter (kg/m²), inclusive, at screening
* Have blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results that are acceptable for the study
* Have had no episodes of severe hypoglycemia in the past 6 months (requiring assistance in treatment by a second party)
* Have venous access sufficient to allow for blood sampling
* Have provided written consent and are willing to follow study procedures and commit to the study duration

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days from a clinical trial or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have or used to have health problems, laboratory test results, blood pressure or ECG readings that, in the opinion of the doctor, could make it unsafe to participate in the study
* Had blood loss of more than 500 milliliters (mL) within the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area under the Concentration Curve (AUC) of Insulin Lispro | Time 0 to 5 hours post dose on Day 1 and Day 3 of each study period
  PK: AUC of Insulin Lispro

SECONDARY OUTCOMES:
Pharmacodynamics (PD): AUC of Glucose Following a Meal | Time 0 to 5 hours post meal on Day 1 and Day 3 of each of study period
  PD: AUC of Glucose Following a Meal

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company